CLINICAL TRIAL: NCT00743340
Title: A Rollover Protocol to Provide Subjects Completing the FTC-203 Study in South Africa With Continued Access to Emtricitabine
Brief Title: Rollover Study Protocol for Pediatric Patients in South Africa for Continued Access to Emtricitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GS-US-162-0112
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infection; emtricitabine; pediatrics; pediatric patients
MeSH Terms: interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emtricitabine (Experimental): Participants will receive emtricitabine for as long as they continue to meet specific virologic criteria and until either: (1) the participant chooses to discontinue treatment of emtricitabine and withdraw from the rollover protocol; (2) the participant experiences a toxicity that necessitates the permanent discontinuation of emtricitabine, or (3) emtricitabine is approved for market distribution in the participant's country of residence.
  Interventions: Drug: Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine — 6 mg/kg capsule once daily, up to a maximum dose of 200 mg once daily, or 10 mg/mL oral solution once daily, up to a maximum of 240 mg once daily

SUMMARY:
The primary objectives of this trial are to provide FTC-203 study participants in South Africa with continued access to the study drug, emtricitabine (FTC), following completion of the FTC-203 study and to collect long-term safety information in participants receiving emtricitabine in combination with other antiretroviral agents.

ELIGIBILITY:
Key Inclusion Criteria:

* Complete or have previously completed at least through the Week 96 Visit (i.e., 96 weeks on study) for the FTC-203 study.
* Complete all End-of-Study Visit procedures for the FTC-203 study.
* Either (a) have a plasma HIV-1 RNA viral load of ≤ 400 copies/mL at the End-of-Study Visit for the FTC-203 study, or (b) if the subject's plasma HIV-1 RNA viral load at the End-of-Study Visit for FTC-203 study is > 400 copies/mL, their viral load is < 1.0 log10 above the nadir recorded after Week 8 of the FTC-203 study and there is reliable genotypic evidence showing a lack of resistance to emtricitabine.
* A parent or other legal guardian has provided written informed consent to the subject participating in the rollover protocol. As applicable, based on the subject's age and normal institution practice, the subject should additionally provide their written informed consent or assent to participate in the rollover protocol.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2005-11-22 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- South Africa (2):
  - Themba Lethu Clinic, Helen Joseph Hospital, Westdene, Johannesburg
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Soweto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 study sites in South Africa. The first participant was screened on 22 November 2005. The last study visit occurred on 13 February 2017.
Pre-assignment Details: 59 participants were screened.
Groups:
- Emtricitabine: Emtricitabine (FTC) 6 mg/kg capsule once daily, up to a maximum of 200 mg once daily, or 10 mg/mL oral solution once daily, up to a maximum of 240 mg once daily
Period: Overall Study
Arm/Group | Emtricitabine
Started | 50
Completed | 9
Not Completed | 41
Not completed — Study medication non-compliance | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal from the Study | 5
Not completed — Protocol Violation | 1
Not completed — Virologic failure | 8
Not completed — Pregnancy | 1
Not completed — Rolled over to other Gilead Study | 23
Not completed — Participant Relocated | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all enrolled participants who have received at least 1 dose of study drug
Groups:
- Emtricitabine: Emtricitabine 6 mg/kg capsule once daily, up to a maximum of 200 mg once daily, or 10 mg/mL oral solution once daily, up to a maximum of 240 mg once daily
Arm/Group | Emtricitabine
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 49
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Access to, and Received the Intervention
Description: This endpoint has been included to satisfy the requirements of ClinicalTrials.gov. However, there were no prespecified endpoints in this study.
Time Frame: Up to 586 weeks
Population: Participants who were enrolled into the study and received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Emtricitabine
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Time Frame: Up to 586 Weeks + 30 days
Description: * Safety Analysis Set: all enrolled participants who have received at least 1 dose of study drug
  * One participant who resulted in incomplete abortion (System order class: Pregnancy, puerperium and perinatal conditions; Event term: Abortion incomplete) was not counted as part of SAE but was counted under pregnancies.
Arm/Group | Emtricitabine
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Emtricitabine (N=50)
Essential hypertension (Vascular disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 1
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1
Pyrexia (General disorders) | 1
Swelling (General disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Conduct disorder (Psychiatric disorders) | 1
Reactive attachment disorder of infancy or early childhood (Psychiatric disorders) | 1
Breast enlargement (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Appendicitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Post procedural sepsis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT00743340/SAP_000.pdf
  • Study Protocol: Amendment (2013-07-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT00743340/Prot_001.pdf
  • Study Protocol: Original (2005-01-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT00743340/Prot_002.pdf